CLINICAL TRIAL: NCT06496295
Title: Evaluating the Efficacy and Use of the Bouquet Speculum for Cervical Cancer Screening in a Diverse Population of Patients
Brief Title: The Use of a Novel Vaginal Speculum for Cervical Cancer Screening in Sunrise Community Health Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Rocky Vista University, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: IRB #2023-266
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cancer Screening
Keywords: Vaginal Speculum; Cervical Cancer Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Vaginal Speculum Exam — Evaluating the visibility of the cervix, ease-of-use, and comfort of a new vaginal speculum.

SUMMARY:
The specific aim of this research is to determine if the Bouquet Speculum TM , compared to the existing 2-bladed vaginal speculum, provides better visualization of the cervix, is easier for the provider to use and is more comfortable for the patient.

Additionally, the clinician's experience with vaginal speculum exams and the patient's last vaginal speculum exam, parity and self-reported weight classification will be surveyed to see what effect, if any, it has on visualization of the cervix, ease-of use, and comfort level for the patient.

The objective of this project is to investigate the use of a novel, FDA-cleared, 5-petaled vaginal speculum in cervical cancer screening (Pap test and/or HPV probe) on 200 patients from Sunrise Community Health Clinics in the Denver-Metro area.

DETAILED DESCRIPTION:
The Bouquet Speculum TM will be used by a variety of clinicians at Sunrise Clinics including physicians, PAs, and NPs for routine cervical cancer screening including Pap tests and/or HPV probes. 200 women will be selected from the Sunrise Clinics in the Denver-Metro area. Women who do not have a cervix or have never had a vaginal speculum exam will be excluded. The inclusion criteria is women ages 18-65.

The clinician will be provided with a one-page Instructions for Use document and a 2-minute instructional video on how to use the Bouquet Speculum TM. The clinician will then be assigned a letter and complete three questions on a survey for each patient regarding 1. visualization of the cervix 2. ease-of-use 3. experience with speculum exams. The patient will be consented and de-identified and assigned a number to their survey of four questions: 1. comfort level 2. last vaginal speculum exam 3. self-reported description of weight (underweight, normal, overweight, obese) 4. parity (number of births).

The length of the study is anticipated to be three months. The surveys will be collected and tabulated and then evaluated by Dr. Mark Payton who has experience with the Pakistan study.

The Bouquet Speculum has been FDA-cleared and is a Class II medical device and poses a non-significant risk for use in humans.

Proprietary Name: Bouquet Vaginal Speculum Classification Name: RETRACTOR, VAGINAL Product Code: HDL Device Class:2 Regulation Number: 884.4520 Medical Specialty: Obstetrics/Gynecology Registered Establishment Name: Viospex Registered Establishment Number:3012447313 Owner/Operator: Viospex Owner/Operator Number:10051911 Establishment Operations: Manufacture

ELIGIBILITY:
Inclusion Criteria:

* women, gender diverse patients with an intact cervix
* women ages 18-25

Exclusion Criteria: no prior vaginal speculum exam

* under age 18 or over age 65
* lack of a uterine cervix
* no prior vaginal speculum exam

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women, gender diverse patients with an intact cervix
Study Population: Sunrise Community Health Clinics provide affordable health care to the uninsured and underinsured. This particular study involves women or gender diverse patients with a cervix and who have had a previous vaginal speculum exam.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating the use of the Bouquet Speculum for cervical visibility, ease-of-use, and comfort level | 3 months
  200 women will be selected from the Sunrise Clinics in the Denver-Metro area. The clinician will then be assigned a letter and complete three questions on a survey for each patient regarding 1. visualization of the cervix 2. ease-of-use 3. experience with speculum exams. The patient will be consented and de-identified and assigned a number to their survey of four questions: 1. comfort level 2. last vaginal speculum exam 3. self-reported description of weight (underweight, normal, overweight, obese) 4. parity (number of births).
  The Bouquet Speculum has been FDA-cleared and is a Class II medical device and poses a non-significant risk for use in humans. Regulation Number: 884.4520

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bouquet, DO, Principal Investigator — Rocky Vista University
Locations (1):
- Rocky Vista University, Englewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouquet JM, Naji R, Armas CA, Roldan V, Selkhi S, Bentley CZ, Zapata I, Fisher J. An Innovative Design for the Vaginal Speculum. Med Devices (Auckl). 2023 Sep 25;16:211-218. doi: 10.2147/MDER.S415558. eCollection 2023. PMID 37790696
- See also: Publication in the Journal of Women's Health — https://www.longdom.org/open-access/a-new-vaginal-speculum-and-an-inexpensive-kit-to-screen-and-treat-dysplasia-and-cancer-of-the-cervix-44231.html